CLINICAL TRIAL: NCT05607368
Title: Mast Cells Are Involved in the Mechanism of NPSLE Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, HUNAG QIN, Clinical Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: NFEC-2022-005
Record Dates: First submitted 2022-10-26; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SLE group: 1. Voluntary signing of informed consent;
  2. Age greater than 18 years old, less than 50 years old, gender is not limited;
  3. Patients with SLE who meet diagnostic criteria.
- NPSLE epilepsy group: 1. Voluntary signing of informed consent.
  2. Age greater than 18 years old, less than 50 years old, gender is not limited.
  3. Patients with NPSLE epilepsy who meet diagnostic criteria.
- Healthy control group: 1. Voluntary signing of informed consent;
  2. Healthy volunteers older than 18 years old and less than 50 years old, regardless of gender;
  3. No systemic diseases and neurological symptoms and signs;
  4. According to the judge's judgment, healthy volunteers matching the NPSLE epilepsy group in terms of gender, age, and education level were selected as the control group.

SUMMARY:
Tryptase, TLR4, and anti-NR2A antibodies were measured in serum, cerebrospinal fluid, and subjects and other markers to assess their relevance to disease activity, aiming to find new therapeutic targets,Timely intervention to improve the prognosis of SLE and improve the quality of life of patients with SLE.

DETAILED DESCRIPTION:
This study is a prospective cohort study: it is proposed to be divided into 3 groups, namely healthy control group and SLE group, NPSLE epilepsy group; Fifteen cases were included in each group, with the consent of the subjects and signed to know Consent form, record all subjects' clinical and laboratory test data, and test subjects' blood. Markers such as cerebrospinal fluid tryptase, TLR4 and anti-NR2A antibodies, follow-up 2 year, the patient's disease activity is evaluated every year, the change of indicators is dynamically observed, and statistical points are made divide.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy control group

   * Voluntary signing of informed consent;
   * Healthy volunteers older than 18 years old and less than 50 years old, regardless of gender;
   * No systemic diseases or neurological symptoms or signs;
   * According to the judge's judgment, healthy volunteers matching the NPSLE epilepsy group in terms of gender, age, and education level were selected as the control group.
2. SLE group

   * Voluntary signing of informed consent;
   * Age greater than 18 years old, less than 50 years old, gender is not limited;
   * Patients with SLE who meet diagnostic criteria.
3. NPSLE Epilepsy Group

   * Voluntary signing of informed consent;
   * Age greater than 18 years old, less than 50 years old, gender is not limited;
   * Patients with NPSLE epilepsy who meet diagnostic criteria.

Exclusion Criteria:

1. SLE group

   * patients with SLE with other autoimmune diseases;
   * Previous seizures, psychiatric abnormalities and other manifestations;
   * MR of the head has obvious abnormal signals in the skull or EEG shows abnormal signals;
   * History of use of hormones and immunosuppressants;
   * The investigators judged that it was not suitable to participate in this study.
2. NPSLE Epilepsy Group

   * prior history of epilepsy or clear cranial MR findings suggesting structural abnormalities;
   * Presence of precipitating seizures such as sleep deprivation, high fever, infection, long-term abstinence from alcoholism
   * Interrupt, patients with systemic diseases such as hypoglycemia, severe electrolyte disorders, malignant lesions, progressive or degenerative diseases, severe liver and kidney insufficiency and other metabolic diseases;
   * The investigators judged that it was not suitable to participate in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nanfang Hospital presents patients with systemic lupus erythematosus (SLE) and neuropsychiatric lupus(NPSLE) patients with epilepsy, as well as health examinations at the Health Management Center of Southern Hospital Healthy subjects
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in disease activity index | Baseline, months 3, 6, 9, 12, 15, 18, 21, and 24
  SLEDAI
Numerical changes in markers such as tryptase, TLR4, and anti-NR2A antibodies in blood and cerebrospinal fluid | Baseline, months 3, 6, 9, 12, 15, 18, 21, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Qin Huang, Doctor, Principal Investigator — Southern Medical University
Locations (1):
- Qin Huang, Guangzhou, Guangdong, China